CLINICAL TRIAL: NCT02336009
Title: Clinical, Radiological and Patient Perceived Outcome After Total Wrist Arthroplasty With a New Total Wrist Arthroplasty Implant
Brief Title: Patient Perceived Outcome After Total Wrist Arthroplasty With a New Total Wrist Arthroplasty Implant
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Örebro University, Sweden (Other)
Collaborators: Örebro Läns Landsting (Other Government)
Responsible Party: Principal Investigator, Anil Gupta, dr Anil Gupta, MD, FRCA, PhD, Örebro University, Sweden
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Orebro Lans landsting 01-14
Record Dates: First submitted 2014-11-24; First posted 2015-01-12 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Rheumatoid Arthritis; Osteoarthritis
Keywords: wrist arthritis; total wrist arthroplasty
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- total wrist arthroplasty, Trimed (Experimental): This is a pilot study where all patients will be operated with the Trimed total wrist arthroplasty.
  Interventions: Device: total wrist arthroplasty, Trimed

INTERVENTIONS:
Device: total wrist arthroplasty, Trimed — A new total wrist arthroplasty design. A pilot study.

SUMMARY:
Total wrist arthroplasty (TWA) surgery has developed gradually and can offer patients with rheumatoid arthritis/osteoarthritis reduced wrist pain with mainly preserved wrist range of movement. Each year 60-70 patients in Sweden are operated with a total wrist arthroplasty. Several implants are available on the market and they all have different pros and cons. One risk with a total wrist arthroplasty is loosening of the implant. If an implant is loose, revision of the implant to another TWA is sometimes possible, if not, a wrist fusion is the likely alternative. Revision rates five years after the index operation have improved, however, they cannot yet compare with the results after a total hip arthroplasty. A newly designed TWA has been developed by the department of Hand Surgery, Örebro university Hospital, Örebro, Sweden, in cooperation with Trimed Inc. The newly developed TWA offers theoretical advantages and has been biomechanically tested at the Mayo clinic.

This is a pilot study where patients operated with the TWA will be assessed pre and postoperatively according to study protocol in order to evaluate outcome after TWA radiologically, clinically and regarding patient perceived outcome measures.

DETAILED DESCRIPTION:
Method: Patients will be studied preoperatively and after 1, 2, 5, and 10 years with respect to changes of the following outcome measures.

1. Patient related outcome measures: DASH=Disabilities of Arm Shoulder and Hand, COPM=Canadian Occupational Performance Measure, PRWE=Patient Related Wrist Evaluation.
2. Wrist range of motion: dorsal/volar flexion, ulnar/radial deviation, pronation/supination. Hand grip strength, pinch grip, key pinch.
3. Wrist pain. VAS-pain scores (Visual analog score) at rest and in activity.
4. X-ray findings. Implant survival will be studied with Kaplan-Meyer graphs.

ELIGIBILITY:
Inclusion Criteria:

* Painful wrist arthritis
* Wrightington X-ray grade 2-4.

Exclusion Criteria:

* Infection
* Substance abuse
* Mental illness.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-10; Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
revision rate | changes in revision rates up to 10 years postoperatively
  The frequency of TWA implants revised up to 10 years after the index operation

SECONDARY OUTCOMES:
changes in patient related outcome measures (PROM) | 1, 2, 5, and 10 years postoperatively
  Assessed as DASH=Disabilities of Arm Shoulder and Hand, COPM=Canadian Occupational Performance Measure, PRWE=Patient Related Wrist Evaluation preoperatively and after 1, 2, 5, and 10 years postoperatively
Changes in Range of Motion (ROM | 1, 2, 5, and 10 years postoperatively
  flexion, extension, radial and ulnar deviation, pronation, supination. Hand grip strength, pinch grip, lateral grip, and radiographic loosening, VAS-pain scores.

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Pettersson, MD, PhD, Principal Investigator — Orebro County Council, Orebro University
Locations (1):
- Department of Hand Surgery, Örebro, Sweden